CLINICAL TRIAL: NCT03602521
Title: Reactivity of Patients With Borderline Personality Disorder to an Ecological Interpersonal Stress : Pathophysiology of Suicidal Behaviors Study Model
Brief Title: Reactivity of Patients With Borderline Personality Disorder to an Ecological Interpersonal Stress
Acronym: ROI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL17_0394
Record Dates: First submitted 2018-07-18; First posted 2018-07-27 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-06

CONDITIONS: Female; Borderline Personality Disorder
Keywords: Psychiatry; Suicidal Behavior; Borderline Personality Disorder; Interpersonal Relations; Social Stress; Oxytocin; Neuropeptide
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BPD (Experimental): Blood sample After simulating an interpersonal stress, the evolution of plasma neuropeptides level (OXT, vasopressin and opioid) of patients with a BPD
  Interventions: Other: Interpersonal stress
- HC (Active Comparator): Blood sample After simulating an interpersonal stress, the evolution of plasma neuropeptides level (OXT, vasopressin and opioid) of healthy controls (HC) patients .without any history of psychopathology
  Interventions: Other: Interpersonal stress

INTERVENTIONS:
Other: Interpersonal stress — Through an interview the evaluator will make a 1 to 2 pages script, written in first-person and in present tense. It will involve an interpersonal conflict between the participants and the person who once trigger their feeling of abandonment.
  After reading the script the participants will have to close their eyes and imagine the event as if was happening to them, now, in real time, and think about it during 3 minutes.
  To evaluate the stress efficiency, the evaluator will ask 2 questions :
  * 1) "from 0 (no distress at all) to 10 (maximal unimaginable distress), to wich point this script bring distress to you?"
  * 2) "from 0 (I can not at all) to 10 (I can completely), to wich point are you able to imagine the scenario in real time, as if you were living it?"

SUMMARY:
Use lay language.

According to the World Health Organization 1 death by suicide occurs every 40 seconds, leading suicide prevention to one of the public health priority.

BPD (Borderline Personality Disorder) is a common condition affecting 6% of the population.

This disorder is characterized by unstable emotions, unstable mood, difficulties with relationship and feer of abandonment.

Borderline Personality Disorder is also the psychopathology the most related to suicidal attempts.

Indeed, up to 50% of the patients admitted to hospital after a suicide attempt are diagnosis with a Borderline Personality Disorder

Negative interpersonal events (events occurring between two people) are known as the main stressor that trigger a suicidal attempt.

People with a Borderline Personality Disorder are highly sensitive to it.

Moreover, neuropeptides such as oxytocin (OXT), vasopressin and opioid are known to be involved in the regulation of the emotions, especially those linked to relationship.

The purpose of this study is to improve knowledge in suicidal behaviors.

After simulating an interpersonal stress, the evolution of plasma neuropeptides level (OXT, vasopressin and opioid) of patients with a BPD will be compared to healthy controls (HC).

Clinical data reflecting how the participant is feeling will be collected as well.

DETAILED DESCRIPTION:
A dysregulation of the neuropeptides (OXT, vasopressin and opioid) could explain the dysregulation of the emotions of people with Borderline Personality Disorder.

Up to this date there is no other study measuring neuropeptides kinetics of patient with Borderline Personality Disorder after an interpersonal stress.

This task of stress is meant to reproduce what people with Borderline Personality Disorder suffer in their everyday life (ecological).

To reach this point, an imaginary interpersonal stress will be asked to be reproduced by the participants.

Neuropeptides concentrations and clinical data (fear, shame, anger, moral pain, compelling needs (suicidal and non-suicidal)) will be collected at different times (pre stress, post stress immediat, 5 minutes post stress,15 minutes post stress and 40 minutes post stress)

As copeptin ( fragment C terminal of the vasopressin) and vasopressin are found in stoichiometric concentration in the plasma as copeptin is more stable than vasopressin, plasma copeptin level will be used to reflect the one of vasopressin.

The hypothesis is that both the neuropeptide variation and clinical data before and after the interpersonal stress will be higher for the patient with Borderline Personality Disorder than healthy controls.

A correlation between clinical assessments and neuropeptides kinetics is expected. This study will help to identify inter-individual and contextual factors impacting neuropeptide's kinetics

ELIGIBILITY:
Inclusion Criteria:

No specific inclusion criteria :

* If taking hormonal contraceptive: able to participate between the 3rd and 18th day after taking the contraceptive If not taking hormonal contraceptive: able to participate between the 5th and 12th day after the first day of the last period
* Able to understand the nature, purpose and methodology of the study
* Having signed the informed consent
* To be affiliated to a social security scheme

Specific inclusion criteria

Borderline Personality Disorder(BPD) :

- Clinical diagnosis of BPD using the SCID II (Structured Clinical Interview for DSM-IV-TR Axis II Personality Disorders)

Healthy controls:

- No personal history of psychiatric disorders (Axis I ) defined by the MINI International Neuropsychiatric Interview according to the DSM-5 criteria

Exclusion Criteria:

* Refusal of participation
* Subject protected by law (guardianship)
* Life time diagnosis of schizoaffective disorder or schizophrenia
* Pregnant or breastfeeding women
* Deprived of liberty Subject (by judicial or administrative decision)
* Exclusion period in relation to another protocol
* Having reached the maximum annual amount of allowances of € 4,500

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
Variation of plasma oxytocin concentrations after an interpersonal stress | from pre interpersonal stress to 5 minutes post stress
  Evaluate and compare the variation of plasma oxytocin concentrations before and after an interpersonal stress of patients with BPDs vs healthy controls between pre stress to 5 minutes post interpersonal stress.

SECONDARY OUTCOMES:
Evolution of plasma oxytocin concentrations | from pre stress to 40 minutes post interpersonal stress
  Evaluate and compare the evolution of plasma oxytocin concentrations before and after an interpersonal stress of patients with BPDs vs healthy controls. pre stress, post stress immediat, 5 minutes post stress, 15 minutes post stress and 40 minutes post stress.
Evolution of plasma copeptin concentrations | from pre stress to 40 minutes post interpersonal stress
  Evaluate and compare the evolution of plasma copeptin concentrations before and after an interpersonal stress of patients with BPDs vs healthy controls. pre stress, post stress immediat, 5 minutes post stress, 15 minutes post stress and 40 minutes post stress.
Evolution of plasma β-endorphin concentrations | from pre stress to 40 minutes post interpersonal stress
  Evaluate and compare the evolution of plasma β-endorphin concentrations before and after an interpersonal stress of patients with BPDs vs healthy controls. pre stress, post stress immediat, 5 minutes post stress, 15 minutes post stress and 40 minutes post stress.
self-damaging compelling needs(suicidal) pre stress | pre stress before the interpersonal stress
  Basal level of self-damaging compelling needs (suicidal) using a numerical scale (0 = I don't want to kill myself ; 10 = Needs to kill myself maximal imaginable ), before an interpersonal stress.
Evolution of clinical variables: self-damaging compelling needs(suicidal) | from pre stress to 40 minutes post interpersonal stress
  Evolution of the self-damaging compelling needs (suicidal) using a numerical scale (0 = I don't want to kill myself ; 10 = Needs to kill myself maximal imaginable ) post stress immediat, 5 minutes, 15 minutes and 40 minutes after an interpersonal stress of patients with BPDs in comparison to healthy controls.
Evolution of clinical variables: self-damaging compelling needs(non-suicidal) | from post stress immediat to 40 minutes just after the interpersonal stress
  Evolution of the self-damaging compelling needs (suicidal) using a numerical scale (0 = I don't want to kill myself ; 10 = Needs to kill myself maximal imaginable ) post stress immediat, 5 minutes, 15 minutes and 40 minutes after an interpersonal stress of patients with BPDs in comparison to healthy controls..
Clinical variable: self-damaging compelling needs(non-suicidal) | pre stress before the interpersonal stress
  Basal level of self-damaging compelling needs (non-suicidal) using a numerical scale (0 = I don't want to hurt myself ; 10 = Needs to hurt myself maximal imaginable), just before an interpersonal stress.
Evolution of self-damaging compelling needs(non-suicidal) | from post stress immediat to 40 minutes just after the interpersonal stress
  Evolution of the self-damaging compelling needs (non-suicidal) using a numerical scale (0 = I don't want to hurt myself ; 10 = Needs to hurt myself maximal imaginable) post stress immediat, 5 minutes, 15 minutes and 40 minutes after an interpersonal stress, of patients with BPDs in comparison to healthy controls.
psychological pain | pre stress just before the interpersonal stress
  Basal level of psychological pain using a numerical scale (0 =No psychological pain ; 10= Psychological pain maximal imaginable), just before an interpersonal stress.
Evolution of clinical variables: psychological pain | from post stress immediat to 40 minutes just after the interpersonal stress
  Evolution of psychological pain using a numerical scale (0 =No psychological pain ; 10= Psychological pain maximal imaginable) post stress immediat, 5 minutes, 15 minutes and 40 minutes after an interpersonal stress, of patients with BPDs in comparison to healthy controls.
Clinical variable: state of shame | pre stress just before the interpersonal stress
  just before the interpersonal stress Description: Basal level of shame using a numerical scale (0 = No shame ; 10 = Shame maximal imaginable), before an interpersonal stress.
Evolution of clinical variables: state of shame | from post stress immediat to 40 minutes just after the interpersonal stress
  Evolution of the state of shame using a numerical scale (0 = No shame ; 10 = Shame maximal imaginable), post stress immediat, 5 minutes, 15 minutes and 40 minutes after an interpersonal stress of patients with BPDs in comparison to healthy controls.
Clinical variable: state of anger | pre stress just before the interpersonal stress
  Basal level of anger using a numerical scale (0 = No anger ; 10 = Anger maximal imaginable), before an interpersonal stress.
Evolution of clinical variables: state of anger | from post stress immediat to 40 minutes just after the interpersonal stress
  Evolution of the state of anger using a numerical scale(0 = No anger ; 10 = Anger maximal imaginable), post stress immediat, 5 minutes, 15 minutes and 40 minutes after an interpersonal stress of patients with BPDs in comparison to healthy controls
Clinical variable: state of fear | pre stress just before the interpersonal stress
  Basal level of fear using a numerical scale (0 = No fear ; 10 = Fear maximal imaginable), before an interpersonal stress.
Evolution of clinical variables: state of fear | from post stress immediat to 40 minutes just after the interpersonal stress
  Evolution of the state of fear using a numerical scale (0 = No fear ; 10 = Fear maximal imaginable) post stress immediat, 5 minutes, 15 minutes and 40 minutes after an interpersonal stress of patients with BPDs in comparison to healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Ducasse, MD, Principal Investigator — Urgence psychiatric lapeyonie Hospital Montpellier
Locations (1):
- Hospital Lapeyronie, Montpellier, France

IPD SHARING:
Plan to Share IPD: No